CLINICAL TRIAL: NCT03582020
Title: Nutritional Evaluation - NuEva Study
Acronym: NuEva
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Christine Dawczynski,PhD, Head of Junior Research Group Nutritional Concepts, University of Jena
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H8_18
Record Dates: First submitted 2018-06-05; First posted 2018-07-10 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Nutritional Evaluation
Keywords: vegetarians; vegans; flexitarians; western diet
MeSH Terms: interventions — Menu Planning

STUDY DESIGN:
Intervention Model Description: Parallel group design (4 groups), non-randomized Run in (14 d): Food frequency protocol (FFP, 7 d), questionnaires for lifestyle/nutrition/socio-economic status Screening: Fasting blood sample taking, health check Intervention: Four groups differing in their eating habits (pre-condition: stable since at least one year) Intervention - group A: Menu plans for persons who consume a traditional Western diet Intervention - group B: Menu plans for persons who rarely consume meat and meat products (predominantly high-quality products; ≤ 2 times / week) = flexitarians Intervention - group C: Menu plans for vegetarians Intervention - group D: Menu plans for vegans
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Traditional Western Diet (Placebo Comparator): Intervention: Menu plans and recommendations for persons who consume a traditional Western diet (daily consumption of meat and sausage)
  Interventions: Dietary Supplement: menu plans
- Flexitarians (Active Comparator): Intervention: Menu plans and recommendations for persons, who rarely consume meat and meat products (predominantly high-quality products; ≤ 2 times / week) = flexitarians
  Interventions: Dietary Supplement: menu plans
- Vegetarians (Active Comparator): Intervention: Menu plans and recommendations for persons who do not eat meat and sausage (vegetarians)
  Interventions: Dietary Supplement: menu plans
- Vegans (Active Comparator): Intervention: Menu plans and recommendations for persons who do not eat products from animal origin (vegans)
  Interventions: Dietary Supplement: menu plans

INTERVENTIONS:
Dietary Supplement: menu plans — menu plans, recommendations ensuring an optimal nutrient intake according the guidelines of the German Society of Nutrition
  Other Names: menu plans, recommendations

SUMMARY:
The NuEva study focusses on the development and the validation of nutritional concepts for healthy persons with different dietary habits, such as Western diet, flexitarians, vegetarians, as well as vegans. The practical nutritional concepts will ensure an optimal intake of macro- and micronutrients according to the guidelines of the nutritional societies and contribute to prevention and therapy of civilization disease, such as cardiovascular diseases. In addition, the contribution of the nutritional habits on health and disease status (focus cardiovascular diseases) will be evaluated.

DETAILED DESCRIPTION:
The implementation of the vegetarian and vegan lifestyle is characterized by omitting defined food groups such as meat, sausage (vegetarians) or additionally dairy products and honey (vegans). This bears the risk of undersupply with valuable nutrients. Critical nutrients in the vegetarian-vegan lifestyle are low intakes of vitamin B12, vitamin D, n-3 LC-PUFA, calcium, iron, zinc as well as a high phytate intake.

The hype of the vegetarian and vegan lifestyle in combination with hints for critical nutrients following the adoption to these eating habits highlights the need of a comprehensive data collection that allows for making recommendations based on reliable scientific evidence.

To address this need, the proposed NuEva study will enroll 55 vegetarians (adherence of at least 1 year), 55 vegans (adherence of at least 1 year), as well as 55 flexitarians (characteristics: selected and rare meat/sausage consumption, once or twice per week, adherence of at least 1 year). Further, 55 participants who consume a Western diet (adherence of at least 1 year) will be recruited as control group).

Run-in/screening To record and document the varieties in dietary practices within and among each group, the 14 d run-in phase of the proposed study will include individual assessments of dietary habits using self-reports (FFPs, lifestyle questionnaires).

Screening (sampling): comprehensive nutrient analyses (vitamins, minerals, trace elements) in plasma/serum samples

Intervention Based on the screening data, critical nutrients will be identified for each participant and summarized for each group. Based on these data and published scientific data, defined nutrition plans and recommendations ensuring adequate nutrient intake will be developed for each group (according to the guidelines of the German Society of Nutrition (DGE)). The plans are adapted to individual energy requirements based on basal metabolic rate (BMR) and physical activity (PAL) of each study participant. The compliance with the menu plans and the physiological impact on health and disease status will be controlled by analyzing nutrient status in blood samples, which are complemented by metabolomic profiling every 6 months. In addition, a regularly health check and nutritional counselling in combination with the analysis of blood lipids and nutrition status are planned every 3 months. Optionally, we are interested to investigate the relationships between the different dietary habits and the participants' microbiomes. Therefore, collection of feces samples every 12 month is envisaged.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 30 kg/m2
* Participants must be subjectively healthy
* Adherence to one of the four groups (Western diet, flexitarians, vegetarians, vegans) confirmed by lifestyle and nutrition questionnaires, food frequency protocol (7 d)
* Precondition: stable eating habits for at least two years before enrollment

Exclusion Criteria:

* Subjects with any acute or chronic disease (tumor, infection, other), gastrointestinal diseases, diabetes mellitus (type I, II), chronic renal disease, diseases of the parathyroids, diseases necessitating regular phlebotomies
* Intake of additional dietary supplements (e.g. fish oil capsules, vitamins, minerals etc.)
* Weight loss or weight gain (> 3 kg) during the last three months before study begin
* Pregnancy or lactation
* Transfusion of blood in the last three months before blood sample taking

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female (before menopause) and male gender (50 % each)
Enrollment: 55 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
blood lipids after implementation of menu plans | change from baseline after 12, 24, 36 and 48 weeks (optional after 60, 72, 84, 96 weeks)
  LDL/HDL ratio and blood lipids (total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides in mmol/l) after implementation of menu plans

SECONDARY OUTCOMES:
Anthropometric data | change from baseline after 12, 24, 36 and 48 weeks (optional after 60, 72, 84, 96 weeks)
  body mass index (kg/m2)
systolic blood pressure | change from baseline after 12, 24, 36 and 48 weeks (optional after 60, 72, 84, 96 weeks)
  systolic blood pressure (mm Hg)
diastolic blood pressure | change from baseline after 12, 24, 36 and 48 weeks (optional after 60, 72, 84, 96 weeks)
  diastolic blood pressure (mmHg)
Bioelectrical impedance | change from baseline after 12, 24, 36 and 48 weeks (optional after 60, 72, 84, 96 weeks)
  bioelectrical impedance
Basal metabolic rate (BMR) | change from baseline after 48 weeks (optional after 96 weeks)
  basal metabolic rate (BMR)
Fatty acid distribution in plasma lipids und erythrocyte lipids | change from baseline after 48 weeks (optional after 96 weeks)
  Fatty acid distribution in plasma lipids und erythrocyte lipids (> 90 fatty acids, including SFA, MUFA, PUFA; % fatty acid methyl esters (FAME))
vitamin A | change from baseline after 12, 24, 36 and 48 weeks (optional after 60, 72, 84, 96 weeks)
  vitamin A (mmol/l)
vitamin D | change from baseline after 12, 24, 36 and 48 weeks (optional after 60, 72, 84, 96 weeks)
  vitamin D (nmol/l)
vitamin E | change from baseline after 12, 24, 36 and 48 weeks (optional after 60, 72, 84, 96 weeks)
  vitamin E (µmol/l)
vitamin B1 | change from baseline after 12, 24, 36 and 48 weeks (optional after 60, 72, 84, 96 weeks)
  vitamin B1 (nmol/l)
vitamin B6 | change from baseline after 12, 24, 36 and 48 weeks (optional after 60, 72, 84, 96 weeks)
  vitamin B6 (nmol/l)
vitamin B12 | change from baseline after 12, 24, 36 and 48 weeks (optional after 60, 72, 84, 96 weeks)
  vitamin B12 (pmol/l)
folic acid | change from baseline after 12, 24, 36 and 48 weeks (optional after 60, 72, 84, 96 weeks)
  folic acid (µg/l)
calcium | change from baseline after 12, 24, 36 and 48 weeks (optional after 60, 72, 84, 96 weeks)
  calcium (mmol/l)
iron | change from baseline after 12, 24, 36 and 48 weeks (optional after 60, 72, 84, 96 weeks)
  iron (µmol/l)
ferritin | change from baseline after 12, 24, 36 and 48 weeks (optional after 60, 72, 84, 96 weeks)
  ferritin (µg/l)
transferin | change from baseline after 12, 24, 36 and 48 weeks (optional after 60, 72, 84, 96 weeks)
  transferin (g/l)
kalium | change from baseline after 12, 24, 36 and 48 weeks (optional after 60, 72, 84, 96 weeks)
  kalium (mmol/l)
metabolic profiling | change from baseline after 48 weeks (optional after 96 weeks)
  Metabolic profiling (186 endogenous metabolites, AbsoluteIDQ p180 Kit from Biocrates)
high sensitive c-reactive protein | change from baseline after 12, 24, 36 and 48 weeks (optional after 60, 72, 84, 96 weeks)
  high sensitive c-reactive protein (mg/l)
apolipoproteins | change from baseline after 12, 24, 36 and 48 weeks (optional after 60, 72, 84, 96 weeks)
  apolipoprotein AI, B (g/l)
homocysteine | change from baseline after 12, 24, 36 and 48 weeks (optional after 60, 72, 84, 96 weeks)
  homocysteine (µmol/l)
lipoprotein(a) | change from baseline after 12, 24, 36 and 48 weeks (optional after 60, 72, 84, 96 weeks)
  lipoprotein(a) (mg/l)
asymmetric dimethylarginine | change from baseline after 48 weeks (optional after 96 weeks)
  asymmetric dimethylarginine, ADMA (µmol/l)
homoarginine | change from baseline after 48 weeks (optional after 96 weeks)
  homoarginine (µmol/l)
trimethylamine N-oxide | change from baseline after 48 weeks (optional after 96 weeks)
  trimethylamine N-oxide, TMAO (µmol/l)
insulin | change from baseline after 12, 24, 36 and 48 weeks (optional after 60, 72, 84, 96 weeks)
  insulin (mU/l)
HbA1c | change from baseline after 12, 24, 36 and 48 weeks (optional after 60, 72, 84, 96 weeks)
  HbA1c (%)
glucose | change from baseline after 12, 24, 36 and 48 weeks (optional after 60, 72, 84, 96 weeks)
  glucose (mmol/l)
alpha prothrombin time | change from baseline after 12, 24, 36 and 48 weeks (optional after 60, 72, 84, 96 weeks)
  alpha prothrombin time (s)
fibrinogen | change from baseline after 12, 24, 36 and 48 weeks (optional after 60, 72, 84, 96 weeks)
  fibrinogen (g/l)
cystatin C | change from baseline after 48 weeks (optional after 96 weeks)
  cystatin C (marker for kidney function), mg/l
NT-pro-BNP | change from baseline after 48 weeks (optional after 96 weeks)
  NT-pro-BNP (marker for cardiac function, volume regulation), pg/ml
troponin | change from baseline after 48 weeks (optional after 96 weeks)
  troponin (TnT or TnI - marker for myocardial necrosis), pg/ml
galectin 3 | change from baseline after 48 weeks (optional after 96 weeks)
  galectin 3 (marker for fibrosis), ng/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Friedrich-Schiller-University, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: Yes
publication of the study data and results in national and international journals
Supporting Information: Study Protocol
Time Frame: 2021 / 2022
URL: https://www.frontiersin.org/articles/10.3389/fnut.2020.608854/abstract

REFERENCES:
- [Derived] Klein L, Lenz C, Kruger K, Lorkowski S, Kipp K, Dawczynski C. Comparative analysis of fatty acid profiles across omnivorous, flexitarians, vegetarians, and vegans: insights from the NuEva study. Lipids Health Dis. 2025 Apr 9;24(1):133. doi: 10.1186/s12944-025-02517-6. PMID 40205391
- [Derived] Dawczynski C. A Study Protocol for a Parallel-Designed Trial Evaluating the Impact of Plant-Based Diets in Comparison to Animal-Based Diets on Health Status and Prevention of Non-communicable Diseases-The Nutritional Evaluation (NuEva) Study. Front Nutr. 2021 Feb 2;7:608854. doi: 10.3389/fnut.2020.608854. eCollection 2020. PMID 33604351
- See also: Study protocoll (Dawczynski C. A study protocol for a parallel-designed trial evaluating the impact of plant-based diets in comparison to animal-based diets on health and prevention of non-communicable disease - the Nutritional Evaluation (NuEva) study.) — https://www.frontiersin.org/articles/10.3389/fnut.2020.608854/full
- See also: Dawczynski C, Weidauer T, Richert C, Schlattmann P, Dawczynski K, Kiehntopf M. Nutrient intake and nutrition status in vegetarians and vegans in comparison to omnivores - the Nutritional Evaluation (NuEva) study. Frontiers in Nutrition 2022, 9: 819106. — https://www.frontiersin.org/articles/10.3389/fnut.2022.819106/full